CLINICAL TRIAL: NCT04017468
Title: Suprafascial Vancomycin Powder for Prevention of Surgical Site Infections After Instrumented Posterior Spinal Fusion
Acronym: VANCO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital Freiburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-01143
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Active Comparator): The powdered vancomycin will be placed subcutaneously over the closed muscle fascia (suprafascially) at the end of the surgery during wound closure.
  Interventions: Drug: Vancomycin
- Control Arm (No Intervention): The control group receiving only a standard preoperative antimicrobial prophylaxis administered intravenously.

INTERVENTIONS:
Drug: Vancomycin — Patients randomized into the treatment arm will receive 1-2 g of vancomycin powder (Vancocin® i.v.) which will be administered above the closed muscle fascia (suprafascially) before closing the subcutaneous tissue and skin. The dose of the drug will depend on the length of the skin incision: 1 g for incisions ≤ 20 cm, 2 g for incisions ≥ 20 cm.
  Arms: Treatment Arm

SUMMARY:
Surgical site infections (SSI) after spine surgery may occur in up to 12% of cases and can lead to increased morbidity, and healthcare costs In this randomized controlled trial the investigators aim to prospectively investigate the efficacy and safety of suprafascial intrawound vancomycin powder in reducing the rate of SSIs after instrumented spinal fusion surgery. Secondary aims of the study are the incidence of vancomycin-related complications, vancomycin-resistant bacterial infections in the treatment arm as well as the rate of revision surgeries due to SSIs.

DETAILED DESCRIPTION:
Background:

Surgical site infections (SSI) after spine surgery may occur in up to 12% of cases and can lead to increased morbidity, and healthcare costs. Numerous retrospective studies suggest the use of intrawound (subfascial) vancomycin powder in spine surgery to be protective against SSIs. Adverse events, such as seroma formation or neurotoxicity may be associated with the subfascial use of vancomycin powder in high doses in direct proximity to exposed neural structures. Only one retrospective study investigated the use of suprafascial vancomycin powder. The use of intrawound vancomycin powder is controversial and there is a paucity of well-designed prospective trials evaluating its efficacy and safety in spine surgery.

Objective:

The main objective of this Trial is to evaluate the efficacy and safety of suprafascially applied vancomycin powder in open instrumented spine surgery to prevent surgical site infections and inform a future phase-III trial.

Methods:

In addition to standard preoperative systemic antibiotic prophylaxis (SAP), patients in the treatment arm will receive 1-2 g of vancomycin powder (VP) applied above the closed muscle fascia (suprafascial) into the wound at conclusion of the surgery. Patients in the control arm will not receive additional intrawound vancomycin powder. All other intra- and perioperative procedures will be conducted according to standard of practice (SOP) at the respective Trial site. All patient follow-ups and assessment of the surgical site will be observational in nature and adhere to Standard Operating Procedure (SOP) of the Trial site. All patients will be followed up clinically with conventional radiographs after 6 weeks and 3 months after surgery. At each follow-up, clinical assessment and inspection of the surgical site (the wound) will be performed by a blinded assessor (who was not present at index surgery). In cases of evident or suspected SSI standard blood samples and - if required to rule out or confirm a deep SSI - a MRI will be ordered.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age requiring open instrumented dorsal spinal fusion of at least 1 level (involving two adjacent vertebras and one intervertebral disc)
* Signed informed consent

Exclusion Criteria:

* Preoperative ongoing infectious disease present as judged by primary surgeon (based on lab results and clinical assessment);
* Previous spine surgery at index level within last 90 days;
* Known allergy to vancomycin;
* Percutaneous or transmuscular instrumentation (minimally-invasive surgery) only without lumbar interbody fusion;
* Postoperative radiotherapy of surgical site required (e.g. for tumor)
* Preexisting cochlea damage OR known history of hearing loss NOT clearly associated with age-related hearing impairment (presbycusis);
* Renal insufficiency with stage 4 chronic kidney disease (CKD) with a glomerular filtration rate (GFR) of 15-30 ml/min or worse;
* Pregnancy or breastfeeding women;
* Participation in other ongoing clinical trials;
* Patients lacking capacity to consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of superficial and deep SSIs (according to CDC criteria) | within 90 days following index surgery

SECONDARY OUTCOMES:
Rate of revision surgery due to SSIs | within 90 days following index surgery
Rate of vancomycin-resistant bacterial infections in the treatment group | within 90 days following index surgery
Rate of vancomycin-related adverse events both locally and systemically | within 90 days following index surgery
Rate of wound healing disorders without SSI within | within 90 days following index surgery
Rate of wound seromas | within 90 days following index surgery
numeric rating scale (NRS) to assess pain intensity self-reported by the patient (Score 0-10 with 0 representing no pain, and 10 maximum pain intensity) at Visits 3, 4, 5 and 6 for neck or back pain depending on surgical level (cervical or lumbosacral) | day 4, day 5, day 42, day 90
numeric rating scale (NRS) to assess pain intensity self-reported by the patient (Score 0-10 with 0 representing no pain, and 10 maximum pain intensity) at Visits 3, 4, 5 and 6 for leg or arm pain (cervical or lumbosacral) | day 4, day 5, day 42, day 90
Quality of life (EuroQoL 5D-5L), Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/ Depression (rating from no problems to extreme problems) and health status self rating by patient (Score 0-100, 0 the worst health and 100 the best health) | day 42 and day 90
Length of hospital stay | within 90 days following index surgery
Cost of treatment for cost analysis between both treatment arms | 1 year after index surgery
Rate of bony fusion at the level of index surgery as assessed by CT | 1 year after index surgery

CONTACTS AND LOCATIONS:
Overall Officials: Schaer Ralph, MD, Principal Investigator — Inselspital Bern, Department of Neurosurgery
Locations (7):
- Switzerland (7):
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - University Hostpital Bern, Department of Neurosurgery, Bern
  - University Hostpital Bern, Department of orthopaedy, Bern
  - Lindenhofspital Bern, Bern
  - Spitalzentrum Biel, Biel
  - Klinik St. Anna, Lucerne
  - University Hospital Zurich, Department of Neurosurgery, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schar RT, Branca M, Fischer U, Zimmerli S, Soll N. Intrawound vancomycin powder for prevention of surgical site infections after open instrumented posterior spinal fusion (VANCO Trial)-methodology of a randomized, controlled, multicenter study. Trials. 2025 Sep 24;26(1):344. doi: 10.1186/s13063-025-09095-z. PMID 40993807